CLINICAL TRIAL: NCT04802915
Title: Intraoperative Analysis of the Central Retina in Epiretinal Fibrosis
Brief Title: Intraoperative Analysis of the Central Retina in ERF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Collaborators: Makarenko Irina Romanovna (Unknown); Zgoba Mariana Igorevna (Unknown)
Responsible Party: Principal Investigator, Lyskin Pavel Vladimirovich, MD, PhD, MD, PhD, ophthalmosurgeon, The S.N. Fyodorov Eye Microsurgery State Institution
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 124575
Record Dates: First submitted 2020-12-06; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Epiretinal Membrane; Macular Pucker
Keywords: epiretinal membrane; internal limiting membrane; epiretinal fibrosis; macular pucker; central retina
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- epiretinal membrane group (Other): Patient with epiretinal fibrosis confirmed by OCT with BCVA< 0,6 and complaints of metamorphopsies
  Interventions: Procedure: Intraoperative ERM and ILM staining with their assessment and removal

INTERVENTIONS:
Procedure: Intraoperative ERM and ILM staining with their assessment and removal — ERM and ILM staining is performed after vitrectomy. After that we evaluate the condition of macular zone and make a decision to remove the ERM and the need to remove the ILM

SUMMARY:
Changes in the retinal anatomy that occur in epiretinal fibrosis have not been sufficiently studied. It is possible that epiretinal fibrosis leads not only to traction dislocation of the macula, but also to ILM anatomical disorders.

DETAILED DESCRIPTION:
Purpose: to study anatomical changes in the Central retina in epiretinal fibrosis.

Surgical treatment: standard vitrectomy 25-27G; ERM amd ILM stainig by Membrane Blue Dual; epiretinal membrane removal, ILM peeling if the divulsion of ILM was detected.

Expected results: improving the quality of epiretinal fibrosis surgery by obtaining a more detailed picture of the pathological process

ELIGIBILITY:
Inclusion Criteria:

* BCVA < 0,6;

Exclusion Criteria:.

* secondary ERM, glaucoma, diabetic retinopathy, high myopia, BCVA>0,6

Ages: 50 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
ILM integrity | intraoperative
  Visual intraoperative assessment of the ILM integrity
Length and localization of the ILM dialysis | intraoperative
  Length (in degrees) and localization of the ILM dyalisis
ILM displacement | intraoperative
  ILM displacement direction during the formation of detachment and divulsion.
Occurence of ILM dyalisis | intraoperative
  Determination of the ratio of patients with ILM dialysis to the total number of patients with ERF

CONTACTS AND LOCATIONS:
Overall Officials: Pavel V Lyskin, PhD, Principal Investigator — The S.N. Fyodorov Eye Microsurgery State Institution
Locations (1):
- S.N. Fedorov Nmrc "Mntk "Eye Microsurgery", Moscow, Russia

IPD SHARING:
Plan to Share IPD: No